CLINICAL TRIAL: NCT07128875
Title: Effectiveness of Therapeutic Exercises in Reducing Pain and Disability in Knee Osteoarthritis Patients in Older Adults
Brief Title: Therapeutic Exercises for Pain and Disability in Knee Osteoarthritis
Acronym: OA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: RIPHAH-REC Naimat ullah 01018
Record Dates: First submitted 2025-07-14; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis, Knee Pain, Therapeutic Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Exercise; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Group A Therapeutic Group
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: A triple-blind protocol was implemented. Participants with knee osteoarthritis, treating therapists, and outcome assessors were blinded to group assignments. Sham procedures were used in the control group to mimic the active treatment without therapeutic effect. Blinding integrity was periodically assessed through questionnaires evaluating participants' and assessors' guesses regarding group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + TENS + Hot Pack (Experimental): Participants in this group will receive a structured therapeutic exercise program designed to improve physical function and reduce pain in patients with knee osteoarthritis.
  The session includes:
  Warm-Up (10 min): Light walking or stationary cycling
  Range of Motion (ROM) Exercises: Heel slides, seated knee flexion/extension
  Strengthening Exercises:
  Quadriceps sets
  Straight leg raises
  Mini squats (within pain-free range)
  Seated knee extensions using resistance bands
  Stretching Exercises:
  Hamstring stretch
  Calf stretch
  Quadriceps stretch
  Cool Down (5-10 min): Breathing and relaxation techniques
  Modalities:
  Hot Pack: 15 minutes (applied pre- and post-exercise)
  TENS: 10 minutes (applied pre- and post-exercise using dual-channel portable TENS unit - [Brand/Model, if available])
  Interventions: Other: Exercise + TENS + Hot Pack
- Exercise Only (Control) (Active Comparator): Participants in the control group will follow the same structured therapeutic exercise program as the experimental group. However, TENS will be replaced with a sham procedure that mimics device placement without electrical stimulation.
  Warm-Up (10 min): Light walking or stationary cycling
  Range of Motion (ROM) Exercises: Heel slides, seated knee flexion/extension
  Strengthening Exercises:
  Quadriceps sets
  Straight leg raises
  Mini squats (within pain-free range)
  Seated knee extensions using resistance bands
  Stretching Exercises:
  Hamstring stretch
  Calf stretch
  Quadriceps stretch
  Cool Down (5-10 min): Breathing and relaxation techniques
  Modalities:
  Hot Pack: 15 minutes (if applicable)
  Sham TENS: Electrodes applied without current
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise + TENS + Hot Pack — Therapeutic Exercises with Hot Pack and TENS This intervention focuses on improving physical function and reducing pain through structured therapeutic exercises for knee OA patients. The program includes Warm-Up (10 min): Light walking or stationary cycling. 2. Range of Motion (ROM) Exercises: Heel slides, seated knee flexion/extension. 3. Strengthening Exercises:
  Quadriceps sets Straight leg raises Mini squats (pain-free range)
  Seated knee extensions with resistance band 4. Stretching Exercises:
  Hamstring stretch Calf stretch Quadriceps stretch 5. Cool Down (5-10 min): Breathing and relaxation. 6. Hot Pack (15 min) + TENS (10 min): Applied pre and post exercises for pain relief and muscle relaxation.
  Arms: Exercise + TENS + Hot Pack
Other: Exercise — Warm-Up (10 min): Light walking or stationary cycling. 2. Range of Motion (ROM) Exercises: Heel slides, seated knee flexion/extension. 3. Strengthening Exercises:
  Quadriceps sets Straight leg raises Mini squats (pain-free range)
  Seated knee extensions with resistance band 4. Stretching Exercises:
  Hamstring stretch Calf stretch Quadriceps stretch 5.
  Arms: Exercise Only (Control)

SUMMARY:
This study aims to evaluate the effectiveness of structured therapeutic exercises in reducing pain and disability among older adults diagnosed with knee osteoarthritis. The intervention will involve a supervised physical therapy program targeting muscle strength, joint mobility, and functional capacity. Participants will undergo 6 weeks of therapy, and improvements in pain and physical function will be measured using validated scales.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a leading cause of chronic pain and mobility limitations in the elderly population. Therapeutic exercises play a significant role in managing OA symptoms by strengthening the quadriceps, improving joint flexibility, and reducing stiffness. This study will enroll 60 participants aged 50-75 years diagnosed with knee OA. They will undergo a combination of strengthening, range of motion (ROM), and stretching exercises tailored to their condition. The intervention also includes adjunctive modalities such as hot pack and TENS to reduce pain and facilitate muscle engagement. Outcome measures will assess pain intensity, functional ability, and lower limb endurance before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:Minimum Age: 50 Years Maximum Age: 75 Years Sex: All Accepts Healthy Volunteers: No

Inclusion Criteria:

* Diagnosed with knee OA
* Aged 50-75 years
* Experiencing pain or functional limitation
* Able to attend supervised sessions
* Provided informed consent

Exclusion Criteria:- History of total knee replacement

* Severe cardiovascular or neurological conditions
* Acute injury or fracture in lower limb
* Uncontrolled hypertension or diabetes

Ages: 35 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Estimated)
Dates: Start 2025-08-17 (Estimated); Primary Completion 2026-07-17 (Estimated); Study Completion 2026-07-17 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 6 Months
  Pain intensity will be assessed using the Visual Analog Scale (VAS), which ranges from 0 to 10, where 0 indicates no pain and 10 indicates the worst imaginable pain. Higher scores represent worse outcomes.

SECONDARY OUTCOMES:
Change in Physical Disability | 6months
  Physical disability will be measured using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). The WOMAC consists of 24 items scored from 0 (none) to 4 (extreme), yielding a total score range from 0 to 96, where higher scores indicate worse disability

CONTACTS AND LOCATIONS:
Overall Officials: Dr Nadeem Ahmad, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah international University Malakand Campus, Malakand, Kpk, Pakistan

IPD SHARING:
Plan to Share IPD: No